CLINICAL TRIAL: NCT00579033
Title: Tactile Operant Conditioning To Alleviate Focal Hand Dystonia Symptoms
Brief Title: Somatosensory Processing in Focal Hand Dystonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Dystonia Medical Research Foundation (Other)
Responsible Party: Aimee Nelson, Assistant Professor, Toronto Western Research Institute, University of Waterloo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05-0959-A; 05-0959-A
Record Dates: First submitted 2007-12-17; First posted 2007-12-21 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-03

CONDITIONS: Focal Hand Dystonia; Musician's Dystonia; Writer's Cramp; Dystonic Cramp
Keywords: somatosensory; cortex; neuroimaging; tactile; cortical plasticity; dystonia
MeSH Terms: conditions — Dystonia, Focal, Task-Specific; Dystonic Disorders; Dystonia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Sham Comparator)
  Interventions: Other: Tactile training + sham rTMS
- 2 (Active Comparator)
  Interventions: Other: Tactile training + rTMS

INTERVENTIONS:
Other: Tactile training + sham rTMS — tactile training for 2.5/hr/day for 15 days - this plus the sham rTMS
  Arms: 1
Other: Tactile training + rTMS — tactile training 2.5/hr/day for 15 days plus daily 5Hz rTMS
  Arms: 2

SUMMARY:
Patients with focal dystonia experience uncontrollable movements of the hand during certain types of skilled movements. Though the origin of the disorder is not fully understood, it is thought that brain areas involved in moving the hands and receiving touch information from the hands, are involved. For example, patients with dystonia affecting the hand show changes in their ability to perceive touch - this is something that typically escapes the patients own awareness. Further, the area of the brain receiving touch information has a disrupted representation of the finger skin surfaces.

The goal of our research is to improve dystonia symptoms in patients with hand dystonia. We will attempt to achieve this goal by implementing an intensive training treatment that requires patients to attend to, and use touch information applied to specific fingertips. Previous work has attempted to alter touch perception using sensory training and improvements in motor control (hand writing) of dystonia patients were observed. For example, learning to read Braille improves tactile perception and handwriting in focal hand dystonia. A different approach to treat focal hand dystonia involves a technique called repetitive transcranial magnetic stimulation (rTMS), and this can also temporarily improve hand writing in dystonia patients. The proposed research will attempt to alter touch processing using touch training alone, or in combination with rTMS. Rather than train using Braille reading, the sensory training will be applied using a systematic, experimenter controlled stimulus set that focuses on touch stimuli applied to individual digits. Importantly patients will have to associate certain types of touch information with rewards and other touch input with the lack of a reward.

The study will first involve measuring the location and representation of the touch in the brain using multiple brain mapping tools. These tools include functional magnetic resonance imaging and magnetoencephalography; when both tools are used a very accurate picture of finger representation can be obtained, and we also know what brain areas respond to touch stimuli. Dystonia symptoms and touch perception will also be assessed. Next, patients will participate in a training intervention that involves 15 days(2.5 hr/day) of touch training applied to the fingertips of the dystonia affected hand. Patients will identify the touch targets amongst distractors and receive on-line performance feedback. The goal of the training is to provide the cortex with regular boundaries of fingers and in this way, attempt to re-shape the sensory cortex to accept these boundaries. Another group of patients will receive rTMS. The goal of the rTMS is to create an environment in sensory cortex that is open or 'ready' to accept changes induced by tactile stimulation. The rTMS will be immediately followed by the tactile training. A third group of patients will receive a placebo version of rTMS followed by tactile training. The latter group will allow us to understand if rTMS has a definite effect on the physiology of the patient. Following the 15-day training, we will assess the brains representation of fingertips, changes in dystonia symptoms and changes in the perception of touch stimuli.

This research will advance the treatment of focal hand dystonia and assist the design of precise remediation training tailored to the dystonia patient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of focal hand dystonia including any but not limited to the following:

  * Writer's cramp,
  * Musician's cramp,
  * Dystonic cramp.

Exclusion Criteria:

* Other neurological conditions
* Epilepsy
* Carpal tunnel or disorders of peripheral nerves
* Psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2007-05; Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Dystonia Rating Scale | 4 weeks

SECONDARY OUTCOMES:
Neuroimaging maps of digit representation | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aimee J Nelson, PhD, Principal Investigator — Toronto Western Research Institute, University of Waterloo
Locations (1):
- Toronto Western Hosptial, Toronto, Ontario, Canada